CLINICAL TRIAL: NCT04975880
Title: A Prospective, Multi-Center, Open-Label Assessment of Efficacy and Safety of Quanta SC+ for Home Hemodialysis
Brief Title: Quanta Home Run Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Dialysis Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-001
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Renal Failure
Keywords: Hemodialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Intervention Model Description: Following enrollment participants will begin hemodialysis treatments on the SC+ machine on a prescription of four-hour treatments, three times per week or per facility standard for training within a hemodialysis facility for a minimum of 4 weeks.
  During this time, both patients and caregivers will undergo extensive training and competency sign off on all aspects of safely administering hemodialysis treatment in the home. This 4 week period can be extended week by week to a maximum of 8 weeks until competency sign off is achieved.
  Upon completion of training, a 1 week transition period will occur followed by the home hemodialysis phase (test phase) which consists of 8 weeks of treatments performed 4 times per week, 3.5 hours each treatment in the participant's home setting by the participant or their care partner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hemodialysis Treatments (Other): All subjects will receive hemodialysis treatments using the SC+ machine for all phases of the trial including in-clinic training, transition, and in the home setting.
  Interventions: Device: SC+ Hemodialysis System

INTERVENTIONS:
Device: SC+ Hemodialysis System — Following the in-clinic training phase and one week transition, the intervention of self or care partner hemodialysis delivered in the home setting will occur for 8 weeks.

SUMMARY:
The purpose of this study is to determine non-inferiority in safety and efficacy when Quanta SC+ is used in the self-care home environment compared to a hemodialysis facility.

DETAILED DESCRIPTION:
This clinical trial is being conducted to evaluate the Quanta SC+ hemodialysis System for home use by patients with established kidney failure. A dialysis prescription of 3 sessions per week, 4 hours per session, or facility standard will be provided during the in-clinic training period, followed by the home period with a dialysis prescription of 4 sessions per week, 3.5 hours per session.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of a written informed consent form signed by the participant
2. Age between 18 and 80 years at time of enrollment
3. A care partner must be available for training on SC+ and to be present in the home during all home hemodialysis sessions
4. Participants should be either receiving regular, facility-based hemodialysis therapy for at least 90 days, or in the case of peritoneal patients transitioning to hemodialysis, at least 90 days, or performing home dialysis (with any frequency) for at least 90 days and willing to return to facility for purpose of study, and should be clinically stable and deemed suitable for home dialysis in the opinion of the principal investigator
5. Willing to accept a dialysis prescription of 3 sessions per week, 4 hours each session or facility standard during in-clinic visits; 4 sessions, 3.5 hours each session during in-home sessions
6. In the opinion of the Investigator, participant has well-functioning and stable vascular access (tunneled, central venous catheter, arteriovenous fistula, or graft) that allows a blood flow of at least 300 ml/min
7. Home environment is adequate to ensure that appropriate electrical connections and water supply necessary for the use and storage of the device as assessed by Quanta prior to subject C1 visit. Also ensure that cellular signal and/or WIFI capacity is adequate.
8. Participant or care partner are capable of understanding the nature of procedures and requirements of the study protocol and of home-based hemodialysis, and are willing and capable of complying with protocol and returning to treatment center as stated in protocol
9. Participant or care partner are capable of being trained to use the machine and troubleshoot should an alarm situation occur
10. In the opinion of the treating physician, the subject is able to participate in the trial in terms of social factors and personal functioning
11. Acceptable physical ability of the participant and/or care partner to perform the hemodialysis treatment at home
12. Financial coverage for treatment costs by Medicare, Medicaid, private insurance, or other arrangement acceptable to participant

Exclusion Criteria:

1. Pregnant or trying to become pregnant (women of childbearing potential must use medically accepted contraceptive measures)
2. Predicted life expectancy of less than 12 months from first study procedure
3. Major cardiovascular adverse event in the 3 months prior to screening
4. Fluid overload due to intractable ascites secondary to liver cirrhosis
5. Uncontrolled or unstable blood pressure (systolic BP outside the range 90 to 180 mmHg)
6. Unstable coronary artery disease
7. New York Class III or IV heart failure, or ejection fraction less than 30%
8. Participation in other clinical studies that may interfere with the current protocol
9. Known problems with coagulation
10. Active, life-threatening, rheumatologic disease.
11. Hematocrit less than 28% at enrollment
12. Hemoglobin less than 9 g/dL at enrollment
13. Suffering from active severe infection
14. Seroreactive for hepatitis B surface antigen
15. Suffering from active malignancy with expected deteriorating course within 6-12 months
16. History of severe reactions to dialyzer membrane material
17. Expected to receive an organ transplant during the course of the study
18. Have dementia or inability to understand procedures
19. Lack an ability for self-care
20. Are non-adherent to their current dialysis treatments
21. Experience intra-dialytic hypotension defined as a decrease in systolic blood pressure of greater than or equal to 20 mmHg or a decrease in mean arterial pressure of greater than or equal to 10 mmHg provided that the decrease is associated with clinical events (symptoms) and the need for an intervention (ultrafiltration turned off, bolus of fluid) in 3 of 5 previous treatments
22. Is intolerant to heparin
23. Considered in the investigator's opinion to be clinically unstable for any other reason
24. Undergoing outpatient dialysis for the treatment of acute kidney injury (AKI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Komenda, MD, Study Director — Quanta Dialysis Technology; Christopher T Chan, MD, Principal Investigator — University of Toronto
Locations (13):
- United States (13):
  - Capital Nephrology Medical Group, Sacramento, California
  - Home Dialysis Therapies of San Diego / UCSD, San Diego, California
  - Satellite WellBound, San Leandro, California
  - Satellite - WellBound, San Mateo, California
  - Satellite - WellBound, Santa Rosa, California
  - High Desert Nephrology Medical Group, Victorville, California
  - Ocala RKCHD At Home, Ocala, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - DaVita Home Dialysis of Indianapolis, Indianapolis, Indiana
  - New Hyde Park Dialysis Center, New Hyde Park, New York
  - Hypertension & Kidney Specialists, Lancaster, Pennsylvania
  - aQua Research Institute, LLC, Houston, Texas
  - Northwest Kidney Centers, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants withdrew consent prior to beginning the clinic phase.
Groups:
- Hemodialysis Treatments: All subjects will receive hemodialysis treatments using the SC+ machine for all phases of the trial including in-clinic training, transition, and in the home setting.
  SC+ Hemodialysis System: Following the in-clinic training phase (lasting 4 to 8 weeks) and one week transition, the intervention of self or care partner hemodialysis delivered in the home setting will occur for 8 weeks.
Period: Clinic Training Phase
Arm/Group | Hemodialysis Treatments
Started | 43
Evaluable Population | 35
Completed | 35
Not Completed | 8
Period: Transition Phase
Arm/Group | Hemodialysis Treatments
Started | 35
Evaluable Population | 35
Completed | 35
Not Completed | 0
Period: Home Hemodialysis Phase
Arm/Group | Hemodialysis Treatments
Started | 35
Evaluable Population | 34
Completed | 31
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Evaluable Population: The Evaluable Population was defined as those participants who completed at least 75% of the treatments required by the protocol. The Evaluable Population of this study was 34 participants.
Arm/Group | Evaluable Population
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 10
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34
Vascular Access Type [Count of Participants; unit: Participants]
  Fistula | 19
  Central Line | 9
  Graft | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Standardized Weekly Kt/V (Efficacy)
Description: The primary effectiveness endpoint was the delivery of a mean standardized weekly Kt/V of greater than or equal to 2.1 in both the clinic phase and the home phase. The weekly standard Kt/V is used to assess dialysis effectiveness by taking into account the clearance provided by individual treatments and the number of times per week the participant treated. The weekly standardized Kt/V is calculated using K (clearance of urea), T (treatment time), and V (urea distribution volume). Current practice guidelines include achieving a minimum result of 2.1 with a target of achieving 2.3, with higher values representing better outcomes. A theoretical range for the minimum and maximum standardized weekly Kt/V does not exist.
Time Frame: 4-8 weeks in the clinic training phase and 8 weeks during the home phase.
Measure: Least Squares Mean (Standard Deviation); unit: Kt/V
Groups:
- Clinic Training Phase: Clinic personnel administered treatments while training the participant and caregiver in a clinic setting with a prescription of 3 treatments per week, 4 hours per treatment, using the SC+ machine.
- Home Hemodialysis Phase: Participants and caregivers administered treatments in the home with a prescription of 4 treatments per week, 3.5 hours for each treatment.
Arm/Group | Clinic Training Phase | Home Hemodialysis Phase
Number analyzed (Participants) | 34 | 34
Kt/V | 2.4 (0.04) | 3.0 (0.03)

2. Primary Outcome: Adverse Event Rate
Description: Adverse event rate: the number of adverse events per 100 treatments that occurred during the study, as defined by:
  * Serious adverse event (SAE)
  * Allergic reaction: type A, anaphylactoid or type B dialyzer reactions to dialyzer, blood tubing, or chemical disinfectant.
  * Blood loss: resulting in hemodynamic compromise that led to death, transfusion, or fluid resuscitation with greater than 1 liter of crystalloid IV fluids.
  * Hemolytic reaction: due to disinfectant exposure, dialysate temperature, mechanical failure, or other device related causes.
  * Infection: related to hemodialysis catheter, its tunnel or exit site, arteriovenous fistula (AVF), or arteriovenous graft (AVG).
  * Intradialytic event: a significant clinical event such as loss of consciousness, cardiac arrest, or seizure caused by device failure.
  * Vascular access complication
  * Pyrogenic reaction
Time Frame: 4-8 weeks in the clinic training phase and 8 weeks during the home phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per 100 treatments
Arm/Group | Clinic Training Phase | Home Hemodialysis Phase
Number analyzed (Participants) | 34 | 34
Events per 100 treatments | 6.3 [3.02 to 9.60] | 5.2 [3.29 to 7.11]

3. Secondary Outcome: Rate of Serious Adverse Events (SAEs) Per 100 Treatments.
Description: Number of SAEs per 100 treatments occurring in the in-clinic portion of the study compared with those occurring in the home portion
Time Frame: 4-8 weeks in the clinic training phase and 8 weeks during the home phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events per 100 treatments
Arm/Group | Clinic Training Phase | Home Hemodialysis Phase
Number analyzed (Participants) | 34 | 34
Events per 100 treatments | 0.6 [0.02 to 1.14] | 0.8 [0.30 to 1.24]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during all phases of the primary study: Clinical training (4-8 weeks), transition phase (1 week), and the Home Hemodialysis Phase (8 weeks). Adverse events were collected for a maximum of 17 weeks.
Description: An independent safety and clinical events committee (SCEC) was created, chartered, and maintained while any adverse events were being collected or participants were receiving study treatment to oversee trial safety.
  Adverse events were collected directly from participants using open-ended questions, through clinic progress notes, and other medical records obtained by research sites.
Groups:
- Transition Phase: Participants and caregivers administered treatments in the home under the supervision of clinic personnel for 1 week.
Arm/Group | Clinic Training Phase | Transition Phase | Home Hemodialysis Phase
All-Cause Mortality (participants affected / at risk) | 1/43 | 0/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 5/43 | 0/35 | 8/35
Other Adverse Events (participants affected / at risk) | 3/43 | 0/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic Training Phase (N=43) | Transition Phase (N=35) | Home Hemodialysis Phase (N=35)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrotal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinic Training Phase (N=43) | Transition Phase (N=35) | Home Hemodialysis Phase (N=35)
Laboratory Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing or presenting trial results, the Principal Investigator is to submit copies of any Proposed Manuscripts to Sponsor at least 60 days in advance of submission. If Sponsor determines that the publication or presentation would be detrimental to its or its affiliates' intellectual property interests, an additional 90 days can be instituted to allow Sponsor to take appropriate steps to protect its or its affiliates' intellectual property interests.

DOCUMENTS (2):
  • Study Protocol (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT04975880/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT04975880/SAP_001.pdf